CLINICAL TRIAL: NCT02885883
Title: Non-invasive Quantification of Atrial Fibrosis by MRI in Atrial Fibrillation
Acronym: QUAFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00285-36; 2011-04 (Other: AP HM)
Record Dates: First submitted 2016-08-23; First posted 2016-09-01 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- a control group (Active Comparator)
  Interventions: Device: MRI 3T
- patients with paroxysmal or persistent AF (Experimental)
  Interventions: Device: MRI 3T
- patients with permanent AF (Experimental)
  Interventions: Device: MRI 3T

INTERVENTIONS:
Device: MRI 3T

SUMMARY:
Three groups of patients will be considered: a control group (n = 10); a group of patients with paroxysmal or persistent AF with AF cryoablation procedure - within this group, MRI will replace CT-scan usually performed in routine before the procedure (n = 15); a group of patients with permanent AF (n = 15). MRI study will include pulmonary veins angiography with gadolinium injection (0.20 mmol/kg), 2D-cine imaging and late-enhancement imaging. A 3D gradient-echo sequence(Flash 3-D) will then be applied 20 minutes after the injection, with the following parameters : echo time 0.98 ms, repetition time 2.53 ms, angle 15°, resolution 2.0x1.3x1.0 mm. T1 map and two T2 sequences will be performed so as to determine LA relaxation times. Argus software will be used for post-treatment imaging. Quantitative data will be expressed in mean ± SD. A comparison of T1 and T2 values in LA will be performed between the three groups. Statistics will be performed with SPSS software in bilateral analysis and a value of p < 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

All persons > 18 years, which have:

gp paroxysmal or persistant FA

1. paroxysmal or persistent FA (under one year),
2. refractory to at least one antiarrhythmic drug therapy
3. eligible for an ablation procedure with cryotherapy
4. the patient may benefit from surveillance. gp permanent FA permanent AF ( defined as chronic arrhythmia after 2 failed attempts to electrical cardioversion and / or more than one year old) , and hospitalized for cardiac reasons or not in different cardiology Timone .

Exclusion Criteria:

* age < 18 years,
* cons -indications to MRI ( claustrophobia, pacemakers and implantable cardiac defibrillators , metal chips intra ocular , valvular mechanical prosthesis ) , allergy to gadolinium ,
* renal impairment ( creatinine clearance <60 mL / min)
* pregnant or nursing ( a pregnancy test must be performed for women of childbearing age at the time of inclusion , the result of this test will be communicated to them .
* the MRI examination takes place three months after the inclusion women of childbearing potential should be placed under effective contraception)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-07; Primary Completion 2015-12-19 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
quantitative measure of atrial fibrosis | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- AP HM, Marseille, France